CLINICAL TRIAL: NCT04144556
Title: The Effects of Nintendo Wii® and Conventional Physical Therapy in Functional Capability and Daily Living Activities in Stroke Patients.
Brief Title: Nintendo Wii® and Physical Therapy in Stroke Patients (NW-SP)
Acronym: NW-SP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, Principal Investigator, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ID0026
Record Dates: First submitted 2019-10-27; First posted 2019-10-30 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Stroke
Keywords: Stroke; virtual reality; physical therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nintendo Wii and conventional physical therapy (Experimental): This group of patients will receive, in addition to the exercise program described below, a virtual rehabilitation program through Nintendo Wii. This program will include upper limb training and lower limb balance training. Participants will choose the games they want to perform the session with. "Wii Fit" (balance games) will be used for the treatment of the lower limbs, and "Wii Sports" (bowling, golf and tennis games) will be used for the treatment of the upper limbs.
  Interventions: Other: Nintendo Wii and conventional physical therapy
- Conventional Physical therapy (Active Comparator): A warm-up period using a stationary bicycle, mobility exercises in supine position, active-assisted/passive kinesiotherapy of the lower and upper limbs, strengthening exercises in sitting position, balance, stability and coordination exercises and walking re-education exercises.
  Interventions: Other: Conventional Physical therapy

INTERVENTIONS:
Other: Nintendo Wii and conventional physical therapy — This group of patients will receive, in addition to the exercise program described below, a virtual rehabilitation program through Nintendo Wii. This program will include upper limb training and lower limb balance training. Participants will choose the games they want to perform the session with. "Wii Fit" (balance games) will be used for the treatment of the lower limbs, and "Wii Sports" (bowling, golf and tennis games) will be used for the treatment of the upper limbs.
  Arms: Nintendo Wii and conventional physical therapy
Other: Conventional Physical therapy — A warm-up period using a stationary bicycle, mobility exercises in supine position, active-assisted/passive kinesiotherapy of the lower and upper limbs, strengthening exercises in sitting position, balance, stability and coordination exercises and walking re-education exercises.
  Arms: Conventional Physical therapy

SUMMARY:
Brief Summary: In the present study a program which combines virtual rehabilitation through Nintendo Wii and conventional physical therapy is applied in stroke patients, evaluating functional capability (TUG), gait and balance (POMA and BBS), motor impairment (FMA), daily living activities (Barthel) and complex activities (FAI).

The hypothesis is that a virtual rehabilitation, through the use of Nintendo Wii®, could be used to improve functionality, gait, balance and living activities of people with chronic physical disabilities in addition to a conventional physical intervention program.

Methods: randomized and controlled clinical study of functional and motor parameters of stroke patients. The subjects will be divided into 2 groups: 1) Nintendo Wii and conventional physical therapy 2) control group which will have conventional physical therapy applied. There will be 2 treatment sessions during 4 weeks, with evaluations before the study and after 4 weeks, which include: functional capability (Timed up and go test), gait and balance performance (Tinetti performance-oriented mobility assessment and Berg balance scale), motor impairment (Fugl-Meyer assessment), daily living activities (Barthel Index) and complex activities (Frenchay activity index).

DETAILED DESCRIPTION:
Introduction. Stroke is one of the most common causes of acquired adult disability. Much of the focus of stroke rehabilitation, in particular, the work of physiotherapists, is focused on recovery of physical independence and functional ability during activities of daily living. Physiotherapy based on conventional therapy has been shown to produce good results in recovery progress after stroke. However, patients tend to find the movements involved in this treatment as difficult and monotonous over time. Virtual rehabilitation is a novel therapeutic intervention based on simulation exercises using virtual reality technology.

Objective. The main objective of the present study was to assess whether a virtual rehabilitation program added to a conventional physical therapy intervention results in greater improvements in functional capability, gait, balance and daily activities compared to conventional physical therapy intervention on its own.

Material and Methods Sample: men and women aged 18 to 80 years having had a first simple stroke Study design. Randomized clinical trial with 2 groups: Group 1. 1) Nintendo Wii and conventional physical therapy 2) control group which will have conventional physical therapy applied.

Evaluations. Clinical interview with anthropometric data. There will be 2 evaluations: at the beginning of the study and at the end of the intervention (at 4 weeks).

In addition, it includes the following evaluation instruments:

* Functional capability: Timed up and go test (TUG)
* Gait and balance performance: Tinetti performance-oriented mobility assessment (POMA) and Berg balance scale (BBS)
* Motor impairment: Fugl-Meyer assessment (FMA)
* Daily living activities: Barthel Index.
* Complex activities: Frenchay activity index (FAI)

ELIGIBILITY:
Inclusion Criteria:

* men and women aged 18 to 80 years
* having had a first simple stroke (ischemic or hemorrhagic) in one cerebral hemisphere
* onset of stroke at least 6 months prior to study inclusion
* have physical limitation in the upper limb and/or lower limb function.

Exclusion Criteria:

* have other morbid neurological conditions
* have hand anesthesia
* show severe cognitive impairment that prevents speaking or understanding both questions and simple instructions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-11-02 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Functional capability: Timed up and go test (TUG) | 4 weeks
  The patient is timed from the moment he/she begins to get up from a chair, walks at a safe and comfortable pace to a line on the floor three meters away, turns and walks towards the chair until he or she sits down again. The subject wears his/her usual footwear and walking aids (cane or walker) if necessary. A faster time indicates better functional performance, indicating a time more than 20 seconds a reduced mobility and, in addition, a score of ≥ 13.5 seconds is used to identify an increased risk of falls.
Gait and balance performance | 4 weeks
  The Tinetti Scale has been designed to evaluate the balance in different positions. It consists of sixteen situations divided into two blocks that require the active participation of the patient. One block assesses gait, in which the subject walks with the examiner first with his usual step, returning with a fast but safe step (using his usual walking aids) with a maximum possible score of 12 points; and the other block assesses balance (in seating, standing and transferring from one to another) with a maximum of 16 points being obtained. The maximum overall score between the two blocks is 28 points.
The Berg Balance Scale (BBS) | 4 weeks
  The Berg Balance Scale (BBS) is a 14-item scale that quantitatively evaluates equilibrium (static and dynamic) and fall risk. The items are scored from 0 to 4; (0 = inability to complete the task; 4 = independent completion of the item). The maximum score is 56 points and the risk of falling limit is 45.

SECONDARY OUTCOMES:
Motor impairment: Fugl-Meyer assessment (FMA) | 4 weeks
  It consists of 33 tasks, divided into 4 parts (shoulder-forearm, wrist, hand, and coordination speed), which performance is used to assess quality of motion, reflex activity, and coordination. Each task is rated on a three-point scale (0 points = cannot perform; 2 points = totally accomplished). The higher the score, the less impairment the subject experiences (maximum score = 66 points).
Daily living activities: Barthel Index. | 4 weeks
  It consists of ten items in which the respective disabilities in the proposed domains are valued from 0 to 10 or from 0 to 15 points. It contains 10 activities of daily living and its maximum score reaches 100 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Gemma V Espí López, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marques-Sule E, Arnal-Gomez A, Buitrago-Jimenez G, Suso-Marti L, Cuenca-Martinez F, Espi-Lopez GV. Effectiveness of Nintendo Wii and Physical Therapy in Functionality, Balance, and Daily Activities in Chronic Stroke Patients. J Am Med Dir Assoc. 2021 May;22(5):1073-1080. doi: 10.1016/j.jamda.2021.01.076. Epub 2021 Feb 24. PMID 33639116